CLINICAL TRIAL: NCT06378996
Title: Arrhythmic Mitral Valve Prolapse Detection Using Long-term Ambulatory Rhythm - A Pilot Study
Brief Title: Arrhythmic Mitral Valve Prolapse Detection Using Long-term Ambulatory Rhythm Monitoring
Acronym: ALARM-PILOT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: S68535
Record Dates: First submitted 2024-04-10; First posted 2024-04-23 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Mitral Valve Prolapse; Ventricular Arrythmia
MeSH Terms: conditions — Mitral Valve Prolapse

STUDY DESIGN:
Intervention Model Description: Prospective, single arm, interventional cohort study including 3 different patient cohorts:
  * Cohort 1: Patients with MVP (not previously known with AMVP) and mild to moderate mitral valve regurgitation
  * Cohort 2: Patients with AMVP and mild to moderate mitral valve regurgitation
  * Cohort 3: Patients with MVP and severe mitral valve regurgitation scheduled for surgical intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 14 day monitoring (Experimental)
  Interventions: Diagnostic Test: 14-day rhythm monitoring

INTERVENTIONS:
Diagnostic Test: 14-day rhythm monitoring — Eligible patients will be monitored during 14 days using the Byteflies patch ambulatory rhythm monitor.

SUMMARY:
Mitral valve prolapse (MVP) affects up to 3% of the general population and a small subset of patients is at risk for ventricular arrhythmias. This subgroup is referred to as AMVP (arrhythmic MVP) and was recently defined using the following criteria: (1) Presence of MVP), (2) Ventricular arrhythmia that is either frequent (≥5% total premature ventricular contraction (PVC) burden on Holter) or complex (non-sustained ventricular tachycardia (nsVT), ventricular tachycardia (VT), or ventricular fibrillation (VF)), and (3) The absence of any other well-defined arrhythmic substrate.

Currently, diagnosis is often based on repeated 24-hour Holter monitoring. However, the ventricular arrhythmia burden varies from day-to-day and long-term rhythm monitoring has shown in other pathologies to increase the diagnostic yield with up to 200% (from 22.5% on 24h to 75.3% on 14 days).

This pilot study aims to study the diagnostic yield of long-term rhythm monitoring in patients with MVP as well as the day-to-day variability of ventricular arrhythmias to facilitate power calculation for a future large-scale prospective registry.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years or older
* Mitral valve prolapse diagnosed on previous echocardiography or cardiac MRI
* New York Heart association classification ≥3 for cohort 3 and classification 1 or 2 for cohorts 1 and 2
* Willing and able to provide signed written informed consent
* No contra-indication for long-term monitoring (known allergy to adhesives)

Exclusion Criteria:

* Prior cardiac surgery, including previous mitral valve intervention
* Prior endovascular mitral valve repair (MitraClip)
* Previous catheter ablation of ventricular arrhythmias
* Patients not in sinus rhythm
* Patients on anti-arrhythmic drugs but betablockers
* Known alternative arrhythmic substrate, for example previous myocardial infarction
* Known allergy to adhesives

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Time to arrhythmic mitral valve prolapse detection | 14 days
  The number of days to reach the detection of arrhythmic mitral valve prolapse, defined as a PVC burden ≥ 5%, nsVT, VT or VF
Number of days with high PVC-burden ≥5% | 14 days
  Number of days with a PVC-burden ≥5%
Number of days with complex ventricular arrhythmia (nsVT, VT, or VF) | 14 days
  Number of days with ≥ 1 nsVT, VT or VF episode
Day-to-day variation in percentage PVC burden | 14 days
  Day-to-day variation of the absolute number of PVC burden in percentage

SECONDARY OUTCOMES:
Association between percentage PVC burden and percentage of late gadolinium enhancement on cardiac MRI | 14 days
  Correlation analysis of two continuous variables. The PVC burden will be calculated as the number of PVCs divided by the total number of heartbeats during the 14 days rhythm monitoring. Percentage of late gadolinium enhancement will be calculated as the ratio of the mass of myocardial tissue with late gadolinium enhancement over the total LV mass on cardiac MRI.
Association between mean number of nsVT episodes per 24hours and percentage of late gadolinium enhancement on cardiac MRI | 14 days
  Correlation analysis of two continuous variables. The mean number of nsVT episodes will be calculated as the average of nsVT episoden per day during the 14 days rhythm monitoring. Percentage of late gadolinium enhancement will be calculated as the ratio of the mass of myocardial tissue with late gadolinium enhancement over the total LV mass on cardiac MRI
Association between percentage PVC burden and global longitudinal strain on transthoracic echocardiography | 14 days
  Correlation analysis of two continuous variables. The PVC burden will be calculated as the number of PVCs divided by the total number of heartbeats during the 14 days rhythm monitoring. Global longitudinal strain will be measured using conventional echocardiography on the 2-chamber, 3-chamber, and 4-chamber apical view.
Association between mean number of nsVT episodes per 24hours and global longitudinal strain on transthoracic echocardiography | 14 days
  Correlation analysis of two continuous variables. Correlation analysis of two continuous variables. The mean number of nsVT episodes will be calculated as the average of nsVT episoden per day during the 14 days rhythm monitoring. Global longitudinal strain will be measured using conventional echocardiography on the 2-chamber, 3-chamber, and 4-chamber apical view.

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No